CLINICAL TRIAL: NCT01148862
Title: An In-clinic, Randomized, Cross-Over Study to Assess the Efficacy of the Low Glucose Suspend (LGS) Feature in the MiniMed Paradigm® X54 System With Hypoglycemic Induction From Exercise
Brief Title: Assess the Efficacy of the Low Glucose Suspend (LGS) Feature in the MiniMed Paradigm® X54 System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CEP235/Z25
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: ASPIRE (Automation to Simulate Pancreatic Insulin Response); X54; Medtronic Diabetes; Diabetes Mellitus; Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Other): Group A will wear the MiniMed Paradigm® X54 System with the Low Glucose Suspend (LGS) feature activated
  Interventions: Device: The MiniMed Paradigm® X54 System
- Group B (Other): Group B will wear the MiniMed Paradigm® X54 System with the Low Glucose Suspend (LGS) feature deactivated
  Interventions: Device: The MiniMed Paradigm® X54 System

INTERVENTIONS:
Device: The MiniMed Paradigm® X54 System — The MiniMed Paradigm® X54 System: A insulin pump equipped with a number of features to actively manage the user's glucose levels. One example is the "Low Glucose Suspend (LGS)" feature. The LGS feature is only available when the pump is used with the subcutaneous glucose sensor for continuous glucose monitoring. To use this feature, the user will be required to select a sensor low suspend limit, or threshold, at which the LGS feature will be triggered. When this feature is selected, if the sensor glucose reading reaches the level that is equal to or less than the programmed threshold, the user receives an alert and the pump suspends.
  Other Names: MiniMed Paradigm® X54 Pump (X54 Pump)

SUMMARY:
The purpose of this study is to assess the efficacy of the Low Glucose Suspend (LGS) feature in reducing hypoglycemia with the MiniMed Paradigm® X54 System with hypoglycemic induction from exercise.

The study will consist of a total of 50 subjects, age 16 through 60 years with Type 1 Diabetes Mellitus.

DETAILED DESCRIPTION:
50 subjects with previously diagnosed Type 1 Diabetes Mellitus will be studied. The subject population includes the following subsets: 4 pediatric subjects aged 16 -17 years, 4 young adult subjects age 18-21 years, and 42 adult subjects age 22-60 years at time of enrollment. Results for all subjects will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between the ages of 16 - 60 years old
* A clinical diagnosis of Type 1 Diabetes Mellitus, as determined by the Investigator, for a minimum of 12 months duration
* Subject has been on a Medtronic insulin pump for at least 3 months, which includes but is not limited to those on sensor augmented insulin pump therapy
* Subject has an A1C value between ≥ 7.0% and ≤ 10.0% at time of enrollment; as measured during the screening visit
* Subject must have a documented stress treadmill test within the last three years of enrollment if the subject had diabetes for >20 years
* Subject willing to follow protocol and procedures for study.

Exclusion Criteria:

* Systolic blood pressure on screening visit is >140 Millimeters of Mercury
* Diastolic blood pressure on screening visit is >90 Millimeters of Mercury
* Subject has a history of hypoglycemic seizure or hypoglycemic coma within the last two years
* Subject unable to tolerate tape adhesive in the area of sensor placement;
* Subject has any active adverse skin condition in the area of sensor placement (i.e. psoriasis, rash, staphylococcus infection) that is not resolved at the time of enrollment
* Subject is pregnant or plans to become pregnant during the course of the study
* Subject has a history of myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack, cerebrovascular accident, angina, congestive heart failure, ventricular rhythm disturbances or thromboembolic disease
* Subject has active Graves disease
* Subject with renal impairment or creatinine above the normal reference range (of the laboratory that the clinical site is utilizing), as demonstrated by the screening laboratory value
* Subject is outside of the normal reference range (of the laboratory that the clinical site is utilizing) for hematocrit, as demonstrated by screening laboratory value
* Subject is outside of the normal reference range (of the laboratory that the clinical site is utilizing) for potassium, as demonstrated by screening laboratory value
* Subject is outside of the normal reference range (of the laboratory that the clinical site is utilizing) for Thyroid-Stimulating Hormone (TSH), as demonstrated by screening laboratory value
* Subject is outside of the normal reference range (of the laboratory that the clinical site is utilizing) for free Thyroxine (T4), as demonstrated by screening laboratory value
* Subject has history of smoking for >5 years
* Electrocardiogram findings observed during the screening visit, which are deemed by the investigator to represent active ischemia or a condition that would compromise subject safety
* The stress treadmill (if subject met inclusion criteria #7) results are deemed by the investigator to represent active ischemia or a condition that would compromise subject safety
* Subject is currently participating in an investigational study (drug or device)
* Subject is currently on beta blocker medication
* Subject has taken oral or injectable steroids within the last 30 days
* Subject is deemed by the Investigator to be unwilling or unable to follow the protocol
* Subject has a history of diagnosed medical eating disorder
* Subject has a history of known illicit drug abuse
* Subject has a history of known abuse with prescription medication
* Subject has a history of visual impairment which would not allow subject to participate in the study and perform all study procedures safely per investigator discretion
* Subject has a history of current alcohol abuse
* Any other condition including abnormalities found on the screening tests which in the opinion of the Investigator, may preclude him/her from participating in the study

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Buckingham, MD, Principal Investigator — Stanford University
Locations (5):
- United States (5):
  - AMCR Institute, Escondido, California
  - Stanford University, Stanford, California
  - Barbara Davis Center of Childhood Diabetes, Aurora, Colorado
  - Barbara Davis Center for Childhood Diabetes, Denver, Colorado
  - Rainier Clinical Research Institute, Renton, Washington

REFERENCES:
- [Derived] Garg S, Brazg RL, Bailey TS, Buckingham BA, Slover RH, Klonoff DC, Shin J, Welsh JB, Kaufman FR. Reduction in duration of hypoglycemia by automatic suspension of insulin delivery: the in-clinic ASPIRE study. Diabetes Technol Ther. 2012 Mar;14(3):205-9. doi: 10.1089/dia.2011.0292. Epub 2012 Feb 8. PMID 22316089

RESULTS

PARTICIPANT FLOW:
Groups:
- LGS on First, Then LGS Off: LGS on first, then LGS off group will wear the MiniMed Paradigm® X54 System with the Low Glucose Suspend (LGS) feature turned 'ON' first, then LGS turned 'OFF' after crossing over
- LGS Off First, Then LGS on: LGS off first, then LGS on group will wear the MiniMed Paradigm® X54 System with Low Glucose Suspend (LGS) turned 'OFF' first, then LGS turned on 'ON' after crossing over
Period: First Intervention
Arm/Group | LGS on First, Then LGS Off | LGS Off First, Then LGS on
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0
Period: Washout Period of 2 Weeks
Arm/Group | LGS on First, Then LGS Off | LGS Off First, Then LGS on
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | LGS on First, Then LGS Off | LGS Off First, Then LGS on
Started | 25 | 25
Completed | 25 | 23
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to LGS on first and LGS off first
Arm/Group | Entire Study Population
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 45
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: The Primary Treatment Comparison is the Evaluation of the Duration (Minutes) of Induced Hypoglycemia.
Description: Duration (minutes) of induced hypoglycemia (YSI < 70 mg/dL)
Time Frame: approximately 8 hours per induction experiment
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- LGS on: Low Glucose Suspend (LGS) Feature Turned 'ON': LGS on: Low Glucose Suspend (LGS) feature turned 'ON'
- LGS Off: Without Low Glucose Suspend (LGS) Feature: LGS off: Without Low Glucose Suspend (LGS) feature
Arm/Group | LGS on: Low Glucose Suspend (LGS) Feature Turned 'ON' | LGS Off: Without Low Glucose Suspend (LGS) Feature
Number analyzed (Participants) | 50 | 50
minutes | 138.5 (76.68) | 170.7 (75.91)
Statistical Analysis 1: Comparison: LGS on: Low Glucose Suspend (LGS) Feature Turned 'ON' vs LGS Off: Without Low Glucose Suspend (LGS) Feature; Test type: Superiority or Other; p = 0.006, ANCOVA; Mean Difference (Final Values) = 32.2

2. Primary Outcome: The Primary Treatment Comparison is the Evaluation of the Severity (Milligrams Per Deciliter) of Induced Hypoglycemia.
Description: Severity (Milligrams per Deciliter) of induced hypoglycemia (YSI < 70 Milligrams per Deciliter) is defined as 70 Milligrams per Deciliter minus absolute lowest blood sugar level
Time Frame: approximately 8 hours per induction experiment
Measure: Mean (Standard Deviation); unit: Milligrams per Deciliter
Arm/Group | LGS on: Low Glucose Suspend (LGS) Feature Turned 'ON' | LGS Off: Without Low Glucose Suspend (LGS) Feature
Number analyzed (Participants) | 50 | 50
Milligrams per Deciliter | 10.5 (5.72) | 12.5 (5.69)
Statistical Analysis 1: Comparison: LGS on: Low Glucose Suspend (LGS) Feature Turned 'ON' vs LGS Off: Without Low Glucose Suspend (LGS) Feature; Test type: Superiority or Other; p = 0.015, ANCOVA; Mean Difference (Final Values) = 2

ADVERSE EVENTS:
Time Frame: Severe adverse event data and adverse event data were collected during the 35-46 days of study duration
Arm/Group | LGS Off: Without Low Glucose Suspend (LGS) Feature | LGS on: Low Glucose Suspend (LGS) Feature Turned 'ON'
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 21/50 | 1/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LGS Off: Without Low Glucose Suspend (LGS) Feature (N=50) | LGS on: Low Glucose Suspend (LGS) Feature Turned 'ON' (N=50)
Dental Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0)
Application Site Bleeding (General disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal Infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Track Infection (Infections and infestations) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (2) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skeletal Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Ketonuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Endodontic procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No